CLINICAL TRIAL: NCT01776632
Title: Promoting Physical Activity in Churchgoing Latinas: Fe en Acción (Faith in Action)
Brief Title: Promoting Physical Activity in Churchgoing Latinas
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: San Diego State University (Other)
Collaborators: National Cancer Institute (NCI) (NIH)
Responsible Party: Principal Investigator, Elva Arredondo, Principal Investigator, San Diego State University
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Prevention
Other Study IDs: R01CA138894 (NIH); R01CA138894-05S1 (NIH); R01CA138894-05S2 (NIH)
Record Dates: First submitted 2012-10-29; First posted 2013-01-28 (Estimated); Results first posted 2019-04-16 (Actual); Last update posted 2021-09-29 (Actual); Status verified 2021-09

CONDITIONS: Chronic Disease
MeSH Terms: conditions — Chronic Disease | interventions — Exercise; Mass Screening

STUDY DESIGN:
Who Masked: Participant, Outcomes Assessor
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- Physical activity (Experimental): Latinas exposed to multi-level Faith in Action intervention promoting physical activity.
  Interventions: Behavioral: Physical activity
- Cancer screening (Active Comparator): Latinas exposed to Faith in Action intervention on cancer screening and prevention.
  Interventions: Behavioral: Cancer screening

INTERVENTIONS:
Behavioral: Physical activity — Promotoras led 6 free physical activity (PA) classes per week (2 walking groups, 2 cardio dance, and 2 strength training) at participating churches randomized to the intervention condition. Classes included prayer, warm-up, moderate-to-vigorous PA, cool-down, followed by discussion of a monthly health handout. Participants received copies of the handouts each month by mail, which promoted healthy PA habits. Promotoras conducted up to 5 motivational interviewing calls with each participant over the 2-year intervention using a guide to evaluate participants' PA engagement, barriers to being active, and solutions to those barriers. Promotoras advocated for changes to the social and built environments of the churches and surrounding neighborhoods in order to promote PA and healthy behaviors.
  Other Names: Faith in Action; Fe en Acción
  Arms: Physical activity
Behavioral: Cancer screening — Promotoras provided a 6-session group-based workshop series on cancer screening and prevention (breast, cervical, colorectal, and skin cancers) at participating churches randomized to the attention-control condition. Participants received informational handouts developed by American Cancer Society and the National Cancer Institute to reinforce learning in addition to lists of local cancer screening resources. Promotoras conducted up to 4 motivational interviewing calls with each participant over the 2-year intervention to encourage screening, help overcome barriers to screening, and provide support for goals.
  Arms: Cancer screening

SUMMARY:
The low prevalence of moderate-to-vigorous physical activity (MVPA) among adult Latinas likely contributes to the high rates of cancer and other chronic diseases in this population. The goals of the current study, based largely upon the core principles of the Social Ecological Model, are to design, implement, and evaluate an innovative multi-level intervention promoting physical activity among churchgoing Latinas.

The evidenced-based intervention targets three "tiers" of environmental influences (i.e., church, immediate neighborhood surrounding the church, and community) on activity, as well as MVPA-related personal factors (i.e.., interpersonal, cultural, and perceived environmental variables). The physical activity intervention will be compared with an attention-control condition providing health education on cancer screening and prevention.

Sixteen churches will be randomly assigned to either the physical activity intervention or the attention-control condition. The primary aim of the study is to determine whether a multi-level intervention will increase MVPA among Latina churchgoers in the intervention condition relative to the attention-control condition.

DETAILED DESCRIPTION:
This two-group randomized controlled trial combines innovative and traditional methods for promoting moderate-to-vigorous physical activity (MVPA) and cancer screening (breast, cervical, colorectal, and skin) among Latinas, and is tested simultaneously in a two-group design. Both interventions lasted two years. The study's primary outcome was min/week of accelerometer-assessed MVPA at baseline (M1) and 12 months (M2) and 24 months (M3) following the start of the intervention.We selected cancer screening as a comparison condition given the relevance of this topic to our target community (i.e., low cervical and colorectal cancer screening rates and follow-up). It was hypothesized that over time, participants in the physical activity condition would engage in significantly higher levels of MVPA, compared to participants in the cancer screening condition. We also expected greater changes in individual-, interpersonal-, and environmental-level correlates of physical activity among participants in the physical activity condition compared to those in the cancer screening condition. Conversely, we expected that participants in the cancer screening condition would engage in higher screening rates compared to those in the physical activity intervention.We anticipated greater changes in individual, interpersonal, and environmental correlates of cancer screening in this condition compared to the physical activity condition.

ELIGIBILITY:
Inclusion Criteria:

* Between the ages of 18-65 years of age
* Latino
* Must be a member of a participating church for at least six months
* Live within 10-15 minutes driving distance from the church
* Able to travel to the church during the week
* Able to attend activities at the church during the week
* Attend church activities (worship or otherwise) at least 4 times a month
* Plan on living in same residence for the next 24 months
* Engage in less than 150 minutes of moderate-to-vigorous physical activity per week

Exclusion Criteria:

* Attendance at other churches participating in the study
* Must not have any conditions limiting ability to be physically active
* Pregnant

Ages: 18 Years to 65 Years | Sex: Female | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 436 (Actual)
Dates: Start 2011-05-11 (Actual); Primary Completion 2015-12-21 (Actual); Study Completion 2015-12-21 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Elva M Arredondo, PhD, Principal Investigator — San Diego State University
Locations (1):
- San Diego State University Research Foundation, San Diego, California, United States

REFERENCES:
- [Background] Arredondo EM, Haughton J, Ayala GX, Slymen DJ, Sallis JF, Burke K, Holub C, Chanson D, Perez LG, Valdivia R, Ryan S, Elder J. Fe en Accion/Faith in Action: Design and implementation of a church-based randomized trial to promote physical activity and cancer screening among churchgoing Latinas. Contemp Clin Trials. 2015 Nov;45(Pt B):404-415. doi: 10.1016/j.cct.2015.09.008. Epub 2015 Sep 8. PMID 26358535
- [Background] Haughton J, Ayala GX, Burke KH, Elder JP, Montanez J, Arredondo EM. Community Health Workers Promoting Physical Activity: Targeting Multiple Levels of the Social Ecological Model. J Ambul Care Manage. 2015 Oct-Dec;38(4):309-20. doi: 10.1097/JAC.0000000000000108. PMID 26280587
- [Background] Beard M, Chuang E, Haughton J, Arredondo EM. Determinants of Implementation Effectiveness in a Physical Activity Program for Church-Going Latinas. Fam Community Health. 2016 Oct-Dec;39(4):225-33. doi: 10.1097/FCH.0000000000000122. PMID 27536927
- [Background] Perez LG, Slymen DJ, Sallis JF, Ayala GX, Elder JP, Arredondo EM. Interactions between individual and perceived environmental factors on Latinas' physical activity. J Public Health (Oxf). 2017 Jun 1;39(2):e10-e18. doi: 10.1093/pubmed/fdw061. PMID 27412175
- [Background] Perez LG, Chavez A, Marquez DX, Soto SC, Haughton J, Arredondo EM. Associations of Acculturation With Self-Report and Objective Physical Activity and Sedentary Behaviors Among Latinas. Health Educ Behav. 2017 Jun;44(3):431-438. doi: 10.1177/1090198116669802. Epub 2016 Sep 27. PMID 27679665
- [Background] Perez LG, Carlson J, Slymen DJ, Patrick K, Kerr J, Godbole S, Elder JP, Ayala GX, Arredondo EM. Does the social environment moderate associations of the built environment with Latinas' objectively-measured neighborhood outdoor physical activity? Prev Med Rep. 2016 Oct 19;4:551-557. doi: 10.1016/j.pmedr.2016.10.006. eCollection 2016 Dec. PMID 27818913
- [Background] Tristao Parra M, Porfirio GJM, Arredondo EM, Atallah AN. Physical Activity Interventions in Faith-Based Organizations: A Systematic Review. Am J Health Promot. 2018 Mar;32(3):677-690. doi: 10.1177/0890117116688107. Epub 2017 Jan 13. PMID 29214856
- [Background] Elder JP, Haughton J, Perez LG, Martinez ME, De la Torre CL, Slymen DJ, Arredondo EM. Promoting cancer screening among churchgoing Latinas: Fe en Accion/faith in action. Health Educ Res. 2017 Apr 1;32(2):163-173. doi: 10.1093/her/cyx033. PMID 28380627
- [Background] Soto SH, Arredondo EM, Haughton J, Shakya H. Leisure-Time Physical Activity and Characteristics of Social Network Support for Exercise Among Latinas. Am J Health Promot. 2018 Feb;32(2):432-439. doi: 10.1177/0890117117699927. Epub 2017 Mar 31. PMID 28359166
- [Background] Perez LG, Elder JP, Haughton J, Martinez ME, Arredondo EM. Socio-demographic Moderators of Associations Between Psychological Factors and Latinas' Breast Cancer Screening Behaviors. J Immigr Minor Health. 2018 Aug;20(4):823-830. doi: 10.1007/s10903-017-0633-1. PMID 28752364
- [Background] Perez LG, Kerr J, Sallis JF, Slymen D, McKenzie TL, Elder JP, Arredondo EM. Perceived Neighborhood Environmental Factors That Maximize the Effectiveness of a Multilevel Intervention Promoting Physical Activity Among Latinas. Am J Health Promot. 2018 Feb;32(2):334-343. doi: 10.1177/0890117117742999. Epub 2017 Nov 22. PMID 29166779
- [Result] Arredondo EM, Elder JP, Haughton J, Slymen DJ, Sallis JF, Perez LG, Serrano N, Parra MT, Valdivia R, Ayala GX. Fe en Accion: Promoting Physical Activity Among Churchgoing Latinas. Am J Public Health. 2017 Jul;107(7):1109-1115. doi: 10.2105/AJPH.2017.303785. Epub 2017 May 18. PMID 28520484
- [Derived] Arredondo EM, Haughton J, Ayala GX, Slymen D, Sallis JF, Perez LG, Serrano N, Ryan S, Valdivia R, Lopez NV, Elder JP. Two-year outcomes of Faith in Action/Fe en Accion: a randomized controlled trial of physical activity promotion in Latinas. Int J Behav Nutr Phys Act. 2022 Jul 30;19(1):97. doi: 10.1186/s12966-022-01329-6. PMID 35907867

RESULTS

PARTICIPANT FLOW:
Groups:
- Cancer Screening: Latinas exposed to Faith in Action intervention on cancer screening and prevention.
  Cancer screening: Promotoras provided a 6-session group-based workshop series on cancer screening and prevention (breast, cervical, colorectal, and skin cancers) at participating churches randomized to the attention-control condition. Participants received informational handouts developed by American Cancer Society and the National Cancer Institute to reinforce learning in addition to lists of local cancer screening resources. Promotoras conducted up to 4 motivational interviewing calls with each participant over the 2-year intervention to encourage screening, help overcome barriers to screening, and provide support for goals. Workshops were hosted at the church and promoted through bulletins and service announcements. Faith components were included throughout the intervention, including prayers before and after each workshop and phone call.
Period: Overall Study
Arm/Group | Physical Activity | Cancer Screening
Started | 217 | 219
Completed | 190 | 190
Not Completed | 27 | 29

BASELINE CHARACTERISTICS:
Groups:
- Physical Activity: Latinas exposed to multi-level Fe en Acción intervention promoting physical activity.
  Physical activity: Promotoras led 6 free physical activity (PA) classes per week (2 walking groups, 2 cardio dance, and 2 strength training) at participating churches randomized to the intervention condition. Classes included prayer, warm-up, moderate-to-vigorous PA, cool-down, followed by discussion of a monthly health handout. Participants received copies of the handouts each month by mail, which promoted healthy PA habits. Promotoras conducted up to 5 motivational interviewing calls with each participant over the 2-year intervention using a guide to evaluate participants' PA engagement, barriers to being active, and solutions to those barriers. Promotoras advocated for changes to the social and built environments of the churches and surrounding neighborhoods in order to promote PA and healthy behaviors.
- Total: Total of all reporting groups
Arm/Group | Physical Activity | Cancer Screening | Total
Number analyzed (Participants) | 217 | 219 | 436
Age, Continuous [Mean (Standard Deviation); unit: years] | 44.5 (9.8) | 44.4 (9.4) | 44.4 (9.6)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 217 | 219 | 436
  Male | 0 | 0 | 0
Race/Ethnicity, Customized [Count of Participants; unit: Participants]
  Hispanic/Latino | 217 | 219 | 436
Region of Enrollment [Number; unit: participants]
  United States | 217 | 219 | 436
Accelerometer-based moderate-to-vigorous physical activity (MVPA) [Mean (Standard Deviation); unit: minutes/week] | 98.8 (61.5) | 107.6 (65.8) | 103.2 (63.8)
Self-report leisure-time MVPA [Mean (Standard Deviation); unit: minutes/week] | 71.2 (121.1) | 64.0 (104.1) | 67.6 (112.8)
BMI [Mean (Standard Deviation); unit: kg/m2] | 30.8 (6.6) | 29.9 (5.8) | 30.3 (6.2)
Waist circumference [Mean (Standard Deviation); unit: cm] | 95.8 (15.0) | 94.1 (14.3) | 94.9 (14.7)

OUTCOME MEASURES:

1. Primary Outcome: Accelerometer-based Moderate-to-vigorous Physical Activity (MVPA)
Description: Change from baseline in moderate-to-vigorous physical activity as assessed by accelerometer
Time Frame: assessed at Baseline, 12 and 24 months following implementation of intervention activities, month 12 reported
Population: A total of 369 participants (183 physical activity condition, 186 cancer screening condition) had valid accelerometer data at 12-month follow-up measures. Those without valid data (unmet wear time, lost device, etc) were not included in the analysis.
Measure: Mean (Standard Deviation); unit: minutes/week
Arm/Group | Physical Activity | Cancer Screening
Number analyzed (Participants) | 183 | 186
minutes/week | 144.4 (117.9) | 129.9 (125.6)
Statistical Analysis 1: Comparison: Physical Activity vs Cancer Screening; Test type: Superiority; p = .03, generalized linear mixed effects; difference of adjusted means = 0.15

2. Primary Outcome: Self-report Leisure-time MVPA
Description: Change from baseline in self-reported leisure-time moderate-to-vigorous physical activity
Time Frame: assessed at Baseline, 12 and 24 months following implementation of intervention activities, month 12 reported
Population: A total of 375 participants (187 physical activity condition, 188 cancer screening condition) had valid self-report leisure-time data at 12-month follow-up measures. Those without valid data (incomplete data, etc) were not included in the analysis.
Measure: Mean (Standard Deviation); unit: minutes/week
Arm/Group | Physical Activity | Cancer Screening
Number analyzed (Participants) | 187 | 188
minutes/week | 138.2 (178.0) | 91.7 (134.4)
Statistical Analysis 1: Comparison: Physical Activity vs Cancer Screening; Test type: Superiority; p = .003, generalized linear mixed effects; difference of adjusted means = 0.39

3. Secondary Outcome: Body Mass Index (BMI)
Description: Change from baseline in body mass index (BMI)
Time Frame: assessed at Baseline, 12 and 24 months following implementation of intervention activities, month 12 reported
Population: A total of 361 participants (178 physical activity condition, 183 cancer screening condition) had valid BMI data at 12-month follow-up measures. Those without valid data (incomplete anthrometric measures, etc) were not included in the analysis.
Measure: Mean (Standard Error); unit: kg/m2
Arm/Group | Physical Activity | Cancer Screening
Number analyzed (Participants) | 178 | 183
kg/m2 | 30.18 (0.14) | 30.60 (0.14)
Statistical Analysis 1: Comparison: Physical Activity vs Cancer Screening; Test type: Superiority; p = .04, mixed effects models; difference of adjusted means = -0.43

4. Secondary Outcome: Waist Circumference
Description: Change from baseline in waist circumference
Time Frame: assessed at Baseline, 12 and 24 months following implementation of intervention activities, month 12 reported
Population: A total of 361 participants (178 physical activity condition, 183 cancer screening condition) had valid waist circumference data at 12-month follow-up measures. Those without valid data (incomplete anthropometrics, etc) were not included in the analysis.
Measure: Mean (Standard Error); unit: cm
Arm/Group | Physical Activity | Cancer Screening
Number analyzed (Participants) | 178 | 183
cm | 95.20 (0.49) | 96.56 (0.54)
Statistical Analysis 1: Comparison: Physical Activity vs Cancer Screening; Test type: Superiority; p = .09, mixed effects models; difference of adjusted means = -1.27

ADVERSE EVENTS:
Time Frame: Baseline to 24 months (2 years)
Arm/Group | Physical Activity | Cancer Screening
All-Cause Mortality (participants affected / at risk) | 1/217 | 0/219
Serious Adverse Events (participants affected / at risk) | 0/217 | 0/219
Other Adverse Events (participants affected / at risk) | 1/217 | 0/219
OTHER ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Physical Activity (N=217) | Cancer Screening (N=219)
broken ankle (Injury, poisoning and procedural complications) | 1 (1) | 0 (0) — Study participant fell and broke ankle during walking group

LIMITATIONS AND CAVEATS:
The current study was implemented with Latina women attending Catholic churches, the findings may not generalize to men, members of other ethnic groups, or Latino groups of other denominations.

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: No